CLINICAL TRIAL: NCT03684551
Title: Improving Community Health Worker Performance by Using a Personalised Feedback Dashboard for Supervision: a Randomised Controlled Trial
Brief Title: Improving Community Health Worker Performance With a Supervision Dashboard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ari Johnson, MD (Other)
Collaborators: Muso, Bamako Mali and San Francisco USA (Unknown); Malaria Research and Training Center, Bamako, Mali (Other); University of California, San Francisco (Other); Harvard Medical School (HMS and HSDM) (Other); Medic Mobile, San Francisco, USA (Unknown); Malian Ministry of Health and Public Hygiene (Unknown)
Responsible Party: Sponsor-Investigator, Ari Johnson, MD, Assistant Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1015-0616
Record Dates: First submitted 2018-09-14; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Community Health Worker Performance
Keywords: Community Health Worker; Health worker supervision; Mali; Randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No dashboard supervision tool (Active Comparator): CHWs received monthly individual supervision from a dedicated CHW supervisor. The supervisory feedback session for CHWs in the control arm was not facilitated by a visual Dashboard tool or any personalised quantitative feedback on quantity, speed, or quality of care. CHW supervisors were instructed to continue providing CHWs in the control arm with feedback informed by patient perspectives and direct observation during the individual supervision visit.
  Interventions: Other: The CHW-led health system; Other: The CHW Supervision model
- Dashboard supervision tool (Experimental): CHWs received monthly individual supervision from a dedicated CHW supervisor. For CHWs randomised to the intervention arm, a visual feedback tool, the CHW Performance Dashboard, was employed during individual supervision, starting in January 2016. During the individual supervisory feedback session, this personalised and relative (to the highest performer) quantitative performance feedback helped orient the discussion of strengths and weaknesses, and allowed the CHW to see quantitatively and visually how his/her performance fared the previous month. The feedback provided to CHWs in the intervention arm, therefore, was both quantitative, informed by the Dashboard, and qualitative, informed by patient perspectives and direct observation of CHW service provision during the individual supervision visit.
  Interventions: Other: The CHW-led health system; Other: The CHW Supervision model; Other: The CHW Performance Dashboard

INTERVENTIONS:
Other: The CHW-led health system — During the study period, all CHWs, regardless of treatment arm, performed proactive case detection, the process of conducting at least two hours per day of door-to-door home visits to proactively identify - through health history inquiry and/or disease diagnostics - patients who need care. For all patients identified, CHWs provided doorstep counselling, evaluation, diagnostics, treatment, referral to appropriate health facilities, and follow-up. CHWs provided care in the community without user fees, and were able to refer patients to the reinforced government primary health centres for care without user fees as well. CHWs were residents of the communities they served, and they were required to be available at home or by phone for consultation at any time.
Other: The CHW Supervision model — CHWs in both study arms received monthly individual supervisory sessions and weekly group supervisory sessions from their dedicated CHW supervisor. An individual monthly session of 360 Supervision included: (i) solicitation of patient perspectives of CHW care; (ii) direct observation of CHW doorstep care; and (iii) a one-on-one feedback discussion with or without the CHW Performance Dashboard depending on treatment arm.
Other: The CHW Performance Dashboard — The CHW Performance Dashboard was a graphic display of a CHW's performance along three indicators defined as follows: (i) "Quantity" of care: the number of homes visited during the month; (ii) "Timeliness" of care: the percentage of sick children under five treated within 24 hours of symptom onset during the month; (iii) "Quality" of care: the percentage of sick children under five treated without protocol error among 23 potential errors during the month. The Dashboard displayed an individual CHW's quantity, timeliness, and quality of care indicators from the previous month, using absolute numbers, percentages, and visual graphics, alongside those of the highest performing CHW. During the individual supervisory feedback session, this personalised and relative (to the highest performer) quantitative performance feedback helped orient the discussion of strengths and weaknesses, and allowed the CHW to see quantitatively and visually how his/her performance fared the previous month.
  Arms: Dashboard supervision tool

SUMMARY:
Countries across sub-Saharan Africa are scaling up Community Health Worker (CHW) programmes, yet there remains little high-quality research assessing strategies for CHW supervision and performance improvement. This randomised controlled trial aims to determine the effect of a personalised performance dashboard used as a supervision tool on the quantity, speed, and quality of CHW care. This study is a randomised controlled trial in a large health catchment area in peri-urban Mali. One hundred forty-eight CHWs conducting proactive case-finding home visits were randomly allocated to receive individual monthly supervision with or without the CHW Performance Dashboard from January to June 2016. Randomisation was stratified by CHW supervisor, level of CHW experience, and CHW baseline performance for monthly quantity of care (number of household visits). With regression analysis, we used a difference-in-difference model to estimate the effect of the intervention on monthly quantity, timeliness (percentage of children under five treated within 24 hours of symptom onset), and quality (percentage of children under five treated without protocol error) of care over a six-month post-intervention period relative to a three-month pre-intervention period.

ELIGIBILITY:
Inclusion Criteria:

* To be a CHW in the study site at the time of enrolment (n=148)

Exclusion Criteria:

* CHW who pretested the Dashboard tool (n=2)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Quantity of care | 9 months
  The number of proactive case-finding home visits during the month

SECONDARY OUTCOMES:
Timeliness of care | 9 months
  The percentage of sick children under five treated within 24 hours of symptom onset during the month
Quality of care | 9 months
  The percentage of sick children under five treated without protocol error among 23 potential errors during the month

REFERENCES:
- [Derived] Whidden C, Kayentao K, Liu JX, Lee S, Keita Y, Diakite D, Keita A, Diarra S, Edwards J, Yembrick A, Holeman I, Samake S, Plea B, Coumare M, Johnson AD. Improving Community Health Worker performance by using a personalised feedback dashboard for supervision: a randomised controlled trial. J Glob Health. 2018 Dec;8(2):020418. doi: 10.7189/jogh.08.020418. PMID 30333922